CLINICAL TRIAL: NCT04339101
Title: Phase IIa Study of Addition of Itacitinib With Tacrolimus/Sirolimus Regimen for GVHD Prophylaxis in Fludarabine and Melphalan Non-Myeloablative Conditioning Hematopoietic Cell Transplantation for Acute Leukemias, MDS or MF
Brief Title: Itacitinib, Tacrolimus, and Sirolimus for the Prevention of GVHD in Patients With Acute Leukemia, Myelodysplastic Syndrome, or Myelofibrosis Undergoing Reduced Intensity Conditioning Donor Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19576; NCI-2020-01722 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19576 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Acute Leukemia; Hematologic and Lymphocytic Disorder; Myelodysplastic Syndrome; Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Hematologic Diseases; Myelodysplastic Syndromes; Primary Myelofibrosis | interventions — fludarabine; Melphalan; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (itacitinib adipate, tacrolimus, sirolimus) (Experimental): RIC: Patients receive fludarabine via infusion on days -9 to -5 and melphalan on day -4 in the absence of disease progression or unacceptable toxicity.
  ALLOGENEIC HSCT: Patients undergo HSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive itacitinib PO QD beginning on day -3 and continuing until day 100 in the absence of disease progression or unacceptable toxicity. Patients also receive tacrolimus IV or PO and sirolimus PO beginning day -3 and continuing until day 100 with a taper in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fludarabine; Drug: Itacitinib Adipate; Drug: Melphalan; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Drug: Fludarabine — Given via infusion
  Other Names: Fluradosa
Drug: Itacitinib Adipate — Given PO
  Other Names: INCB-039110 Adipate; INCB039110 Adipate
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; rapamycin; SILA 9268A; WY-090217
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase IIa trial studies the side effects of itacitinib when given together with standard treatment (tacrolimus and sirolimus), and to see how well it works in preventing graft-versus-host-disease (GVHD) in patients with acute leukemia, myelodysplastic syndrome or myelofibrosis who are undergoing reduced intensity conditioning donor stem cell transplantation. GVHD is a common complication after donor stem cell transplantation, resulting from donor immune cells recognizing recipients' cells and attacking them. Adding itacitinib to tacrolimus and sirolimus may reduce the risk GVHD and ultimately improve overall outcome and survival after donor stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Following a patient safety lead-in, estimate graft-versus-host disease free relapse free (GRFS) survival at 1- year post allogeneic stem cell transplantation (alloHCT).

SECONDARY OBJECTIVES:

I. Estimate the cumulative incidence of acute graft-versus-host disease (aGVHD) and non-relapse mortality (NRM) at 100-days post-transplant.

II. Estimate the cumulative incidence of chronic GVHD at 1- and 2-years post-transplant.

III. Estimate the probabilities of overall and progression-free survival (OS/PFS) at 1- and 2-years post-transplant.

IV. Estimate rate of infection and development of second malignancies including lymphoproliferative disorders at 1- and 2-years post-transplant.

V. Assess patients' quality of life (QOL) at day 100 and 1 year post alloHCT.

EXPLORATORY OBJECTIVES:

I. Characterize and evaluate hematologic recovery, donor cell engraftment and immune reconstitution by cell count and flow cytometry of lymphocyte subsets.

II. Characterize changes in aGVHD biomarkers (Reg-3alpha, TNF-RI, and ST2) and a composite biomarker panel (IL2Ralpha, TNF-R1, IL-8, and hepatocyte growth factor), JAK-regulated pro-inflammatory cytokines (i.e., IL-6, TNFalpha, CRP, Beta2 Microglobulin, and IFNgamma) and STAT3 phosphorylation (downstream of JAK signaling) over time and by aGVHD status/grade.

OUTLINE:

REDUCED INTENSITY CONDITIONING (RIC): Patients receive fludarabine via infusion on days -9 to -5 and melphalan on day -4 in the absence of disease progression or unacceptable toxicity.

ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANT (HSCT): Patients undergo HSCT on day 0.

GVHD PROPHYLAXIS: Patients receive itacitinib orally (PO) once daily (QD) beginning on day -3 and continuing until day 100 in the absence of disease progression or unacceptable toxicity. Patients also receive tacrolimus intravenously (IV) or PO and sirolimus PO beginning day -3 and continuing until day 100 with a taper in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then periodically for up to 2 years post- transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Performance status: Karnofsky >= 70%
* Patients with neoplastic hematologic disorders with indication of allogeneic transplant according to the standard guidelines as follows:

  * Acute leukemia (AL) in first complete response (CR1) or subsequent complete response (CR) or active disease with bone marrow (BM) blast of < 5%
  * Myelodysplastic syndrome (MDS) with intermediate-2 or high risk per International Prognostic Scoring System (IPSS) or
  * Myelofibrosis; primary or secondary if intermediate-2 or high risk per Dynamic International Prognostic Scoring System (DIPPS)
* All candidates for this study must have a matched related donor (MRD) who is willing to donate BM or peripheral blood stem cells or an 8/8 allele matched unrelated donor (MUD)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated. In case of active disease, evaluation should be done within 15 days)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated. In case of active disease, evaluation should be done within 15 days)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated. In case of active disease, evaluation should be done within 15 days)
* Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated. In case of active disease, evaluation should be done within 15 days)
* Left ventricular ejection fraction (LVEF) >= 50%

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* If able to perform pulmonary function tests: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO) (diffusion capacity) >= 50% of predicted (corrected for hemoglobin). If unable to perform pulmonary function tests: oxygen (O2) saturation > 92% on room air.

  * Note To be performed within 28 days prior to day 1 of protocol therapy
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combination (combo), hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin measurement [RPR])

  * If HCV positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chemotherapy, radiation therapy, biological therapy, and/or immunotherapy within 21 days prior to day 1 of protocol therapy

  * Note: Conditioning regimen within 21 days prior to day 1 of protocol therapy is not considered as an exclusion criterion
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Psychological issues, no appropriate caregivers identified, or non-compliant to medication
* Uncontrolled medical or psychiatric disorders which may preclude patients to undergo clinical studies (Discretion of the attending physician)
* Active diarrhea due to inflammatory bowel disease or malabsorption syndrome
* Clinically significant uncontrolled illness
* Active, uncontrolled systemic infection (bacterial, viral, or fungal) requiring antibiotics
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Diagnosis of Gilbert's disease
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2026-01-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Haris Ali, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus): RIC: Patients receive fludarabine via infusion on days -9 to -5 and melphalan on day -4 in the absence of disease progression or unacceptable toxicity.
  ALLOGENEIC HSCT: Patients undergo HSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive itacitinib PO QD beginning on day -3 and continuing until day 100 in the absence of disease progression or unacceptable toxicity. Patients also receive tacrolimus IV or PO and sirolimus PO beginning day -3 and continuing until day 100 with a taper in the absence of disease progression or unacceptable toxicity.
  Fludarabine: Given via infusion
  Itacitinib Adipate: Given PO
  Melphalan: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Sirolimus: Given PO
  Tacrolimus: Given IV or PO
Period: Overall Study
Arm/Group | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus)
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus)
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 63 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Graft-versus-host Disease Free Relapse Free (GRFS) at 1 Year
Description: GRFS is defined as time from the date of transplantation to the first time of observing following events: grade 3-4 acute graft versus host disease (GVHD), chronic GVHD requiring systemic treatment, relapse, or death, whichever occurs first. Kaplan-Meier curve will be generated for GRFS.
Time Frame: From the date of transplantation to the first time of observing following events: grade 3-4 acute graft versus host disease (GVHD), chronic GVHD requiring systemic treatment, relapse, or death, whichever occurs first, assessed at 1 year post transplant.
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus)
Number analyzed (Participants) | 59
percentage of probability | 56 [41 to 69]

2. Secondary Outcome: Cumulative Incidence of Grade II-IV Acute GVHD
Description: Acute GVHD will be graded and staged according to the Consensus Grading.
Time Frame: From day 0 (date of stem cell infusion) through 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus)
Number analyzed (Participants) | 59
percentage of probability | 4 [1 to 13]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Kaplan-Meier curve will be generated for PFS.
Time Frame: From the date of stem cell infusion to the date of death, disease relapse/progression, or last follow-up, whichever occurs first, assessed at 1 year post transplant
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus)
Number analyzed (Participants) | 59
percentage of probability | 70 [54 to 81]

ADVERSE EVENTS:
Time Frame: Up to 2 years post transplant.
Arm/Group | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus)
All-Cause Mortality (participants affected / at risk) | 14/59
Serious Adverse Events (participants affected / at risk) | 9/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus) (N=59)
E. Faecalis Bactermia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
GI Bleed (Blood and lymphatic system disorders) | 1 (1)
polymicrobial pneumonia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Intermittent (Gastrointestinal disorders) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 2 (2)
Disease progression (General disorders) | 1 (1)
Tractable nausea and Vomiting (General disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Bordetella Parapertussis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Itacitinib Adipate, Tacrolimus, Sirolimus) (N=59)
Acute Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 51 (57)
Febrile neutropenia (Blood and lymphatic system disorders) | 21 (21)
Generalized Rash (Blood and lymphatic system disorders) | 1 (1)
Hematochezia (Blood and lymphatic system disorders) | 1 (1)
Hypogammaglobulinemia (Blood and lymphatic system disorders) | 1 (2)
Intermittent Nosebleeds (Blood and lymphatic system disorders) | 1 (1)
Left Eat Discomfort (Blood and lymphatic system disorders) | 1 (1)
Left hip Pain (Blood and lymphatic system disorders) | 1 (1)
Left hip Swelling (Blood and lymphatic system disorders) | 1 (1)
Lower Extremity Bilateral Edema (Blood and lymphatic system disorders) | 1 (1)
Oropharyngeal Erythema (Blood and lymphatic system disorders) | 1 (1)
Orthostatic Hypertension (Blood and lymphatic system disorders) | 1 (1)
Pain Plantar bilateral Feet (Blood and lymphatic system disorders) | 1 (1)
Right Groin Tenderness (Blood and lymphatic system disorders) | 1 (1)
Runny Nose (Blood and lymphatic system disorders) | 1 (1)
Scant Vaginal Bleeding (Blood and lymphatic system disorders) | 1 (1)
Throat Pain (Blood and lymphatic system disorders) | 1 (1)
Upper Extremity Bilateral Edema (Blood and lymphatic system disorders) | 1 (1)
Vaginal Thrombus (Blood and lymphatic system disorders) | 1 (1)
Xerostomia (Blood and lymphatic system disorders) | 1 (1)
bilateral submandibular swelling (Blood and lymphatic system disorders) | 1 (1)
gi blood loss (Blood and lymphatic system disorders) | 1 (1)
norovirus (Blood and lymphatic system disorders) | 1 (1)
polyuria (Blood and lymphatic system disorders) | 1 (1)
vitamin D deficient (Blood and lymphatic system disorders) | 1 (1)
vitamin D. Deficiency (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 7 (8)
Sinus tachycardia (Cardiac disorders) | 18 (18)
Wide complex tachycardia (Cardiac disorders) | 1 (1)
Chest Congestion (Congenital, familial and genetic disorders) | 1 (1)
blisters bilateral feet (Congenital, familial and genetic disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
ear discomfort (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (3)
Blurred vision (Eye disorders) | 3 (3)
Eye pain (Eye disorders) | 1 (1)
Vision decreased (Eye disorders) | 1 (1)
pale conjunctiva (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 25 (26)
Bloating (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 35 (38)
Diarrhea (Gastrointestinal disorders) | 55 (60)
Dry mouth (Gastrointestinal disorders) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 8 (8)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 3 (3)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 4 (4)
GI GVHD (Gastrointestinal disorders) | 1 (1)
GI mucositis (Gastrointestinal disorders) | 1 (1)
GI toxicity (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (8)
Hearburn (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Indigestion (Gastrointestinal disorders) | 1 (1)
MOUTH ULCERS (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 32 (32)
Nausea (Gastrointestinal disorders) | 52 (60)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 10 (10)
Rectal pain (Gastrointestinal disorders) | 10 (10)
Rectal ulcer (Gastrointestinal disorders) | 1 (1)
Recurrent GI Bleed (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 36 (37)
apthous ulcer (Gastrointestinal disorders) | 1 (1)
gingival bleeding (Gastrointestinal disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 4 (4)
hematemesis (Gastrointestinal disorders) | 1 (1)
hematochezia (Gastrointestinal disorders) | 1 (1)
oral lesion (Gastrointestinal disorders) | 1 (1)
tongue lesion (Gastrointestinal disorders) | 1 (1)
Face only (General disorders) | 1 (1)
left wrist (General disorders) | 1 (1)
neck (General disorders) | 1 (1)
upper extremities (General disorders) | 1 (1)
2 Detection (oral swab) (General disorders) | 1 (1)
ADV Viremia (General disorders) | 1 (1)
Abdominal Bloating (General disorders) | 1 (1)
Abdominal Cramping (General disorders) | 3 (3)
Abdominal Discomfort (General disorders) | 1 (1)
Acute GI GVHD (General disorders) | 1 (1)
Acute GVHD skin (General disorders) | 1 (1)
Acute renal insufficiency (General disorders) | 2 (2)
Aphasia (General disorders) | 1 (1)
Apthous ulcers ( oral) (General disorders) | 1 (1)
Bilateral Arm Tingling (General disorders) | 1 (1)
Bilateral Foot Pain (General disorders) | 1 (1)
Bilateral Forearm Macular Rash (General disorders) | 1 (1)
Bilateral Hip Pain (General disorders) | 1 (1)
Bilateral Leg soreness (General disorders) | 1 (1)
Bilateral Lower Extremity Edema (General disorders) | 2 (2)
Bilateral Lower Extremity Tingling (General disorders) | 1 (1)
Bilateral Lower extremity Edema (General disorders) | 1 (1)
Bilateral Upper Extremity tremor (General disorders) | 1 (1)
Bilateral hand sensitivity (General disorders) | 1 (1)
Bleeding from picc Site (General disorders) | 1 (1)
Blister bottom of left foot (General disorders) | 1 (1)
Bone Pain under Spine (General disorders) | 1 (1)
C.Diff Colonization positive (General disorders) | 1 (1)
COV-2 Positive (General disorders) | 1 (1)
Candida Albicans, Few Saccharomyces Cervisiae, Buddign yeast spores (General disorders) | 1 (1)
Catheter pain (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Chills (General disorders) | 16 (17)
Clostridioides Difficile Positive (General disorders) | 1 (1)
Clostridioides Difficile Toxin B Gene by PCR detected (General disorders) | 1 (1)
Clostridium Difficile Infection (General disorders) | 1 (1)
Congestion (General disorders) | 1 (1)
Coronavirus HKU1 infection (General disorders) | 1 (1)
Diffuse mucosal bleeding (General disorders) | 1 (1)
Discomfort Left posterior base of tongue (General disorders) | 1 (1)
Double blurred Vision (General disorders) | 1 (1)
Dry Cough (General disorders) | 1 (1)
E. Coli Bacteremia (General disorders) | 1 (1)
Ecchymosis Left Cheek (General disorders) | 1 (1)
Edema Bilateral Lower Extremeties (General disorders) | 1 (1)
Edema Bilateral Lower Extremities (General disorders) | 2 (2)
Edema LE's (General disorders) | 2 (2)
Edema Lower extremeties (General disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 7 (8)
Edema trunk (General disorders) | 3 (3)
Epigastric Discomfort (General disorders) | 2 (2)
Eruthema @ PICC line insertion site (General disorders) | 1 (1)
Erytehmatous Rash Bilateral Forearms (General disorders) | 1 (1)
Erythema Bridge of Nose (General disorders) | 1 (1)
Erythema Right Buccal Mucosa (General disorders) | 1 (1)
Erythematous Rash Chest (General disorders) | 1 (1)
Erythematous Rash Neck (General disorders) | 1 (1)
Facial Edema (General disorders) | 1 (1)
Facial Rash (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 45 (48)
Fever (General disorders) | 40 (40)
Flu like symptoms (General disorders) | 1 (1)
GVHD skin (General disorders) | 1 (1)
Generalized Body Ache (General disorders) | 1 (1)
Generalized Body Aches (General disorders) | 2 (2)
Generalized Body aches (General disorders) | 1 (1)
Generalized Pain (General disorders) | 1 (1)
Generalized body pain (General disorders) | 1 (1)
Generalized edema (General disorders) | 2 (2)
Generalized joint pain (General disorders) | 1 (1)
Generalized pain (General disorders) | 2 (2)
Generalized weakness (General disorders) | 1 (1)
Growth of Staph Species Coag Neg (General disorders) | 1 (1)
HHV6 viremia (General disorders) | 1 (1)
Hand pruritis (General disorders) | 1 (1)
Heartburn (General disorders) | 2 (2)
Hemorrhoids (General disorders) | 1 (1)
Hypertrophy Right Buccal Tissue (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Inflammation around exit site of PICC Line (General disorders) | 1 (1)
Intermittent Nausea (General disorders) | 1 (1)
Intermittent Neuropathy left lower extremity (General disorders) | 1 (1)
Intermittent epigastric pain (General disorders) | 1 (1)
Intermittent productive cough (General disorders) | 1 (1)
Intermittent right flank pain (General disorders) | 1 (1)
Itching (General disorders) | 1 (1)
LLQ abdominal pain (General disorders) | 1 (1)
Left Arm Numbness (General disorders) | 1 (1)
Left Hip Pain (musculoskeletal) (General disorders) | 1 (1)
Left Inner Cheek Erythema (General disorders) | 1 (1)
Left Shoulder Pain (General disorders) | 2 (2)
Left Toe Gout Pain (General disorders) | 1 (1)
Left Wrist bone pain (General disorders) | 1 (1)
Left abdominal Discomfort (General disorders) | 1 (1)
Left shin Injury (General disorders) | 1 (1)
Leg cramping (General disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Lesion Tip of Tongue (General disorders) | 1 (1)
Light Pseudomonas aeruginosa infection (General disorders) | 1 (1)
Lip Tremor (General disorders) | 1 (1)
Lip ulcer (General disorders) | 1 (1)
Liver GVHD (General disorders) | 1 (1)
Lower Extremity Cramps (General disorders) | 1 (1)
Lower Lip lesion (General disorders) | 1 (1)
Lower extremity bilateral pain (General disorders) | 1 (1)
Maculopapular rash scalp (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Neck Itching (General disorders) | 1 (1)
Neck Rash (General disorders) | 1 (1)
Neck Stiffness (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Non Blanchable redness to foot (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 8 (8)
Odynophagia (General disorders) | 1 (1)
Onset Facial Rash (General disorders) | 1 (1)
Oral sensitivity (General disorders) | 1 (1)
Orthostatic Hypotension (General disorders) | 1 (1)
Pain (General disorders) | 11 (14)
Pain ( ears/nose) (General disorders) | 1 (1)
Pain (epigastric) (General disorders) | 1 (1)
Pain (penile) (General disorders) | 1 (1)
Pain LE's (General disorders) | 1 (1)
Pain after CVP insertion (General disorders) | 1 (1)
Paresthesia Toes (General disorders) | 1 (1)
Perianal Discomfort (General disorders) | 1 (1)
Perirectal pain (General disorders) | 1 (1)
Petichial Rash Bilateral Lower Extremity (General disorders) | 1 (1)
Rare Saccharomyces cervisiae (General disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Rash around Edges of PICC line dressing (General disorders) | 1 (1)
Rectal Discomfort (General disorders) | 1 (1)
Relapsed AML (General disorders) | 1 (1)
Rhinitis (General disorders) | 1 (1)
Right Arm Swelling (General disorders) | 1 (1)
Right Flank Pain (General disorders) | 1 (1)
Right Lower Lip Swelling (General disorders) | 1 (1)
Right Sided Abdominal pain (General disorders) | 1 (1)
Right Sided Chest Pain (General disorders) | 1 (1)
Right Sided Jaw Pain (General disorders) | 1 (1)
Right Testicle Edema (General disorders) | 1 (1)
Right lower lip lesions (General disorders) | 1 (1)
Right shoulder Pain (General disorders) | 1 (1)
Right upper extremity Swelling (General disorders) | 1 (1)
Rosacea (General disorders) | 1 (1)
Sciatica pain (General disorders) | 1 (1)
Septic Shock (General disorders) | 1 (1)
Shoulder pain (General disorders) | 1 (1)
Sore gums (General disorders) | 1 (1)
Spasm and tingling of right hand (General disorders) | 1 (1)
Stomach pain (General disorders) | 1 (1)
Stress incontinence (General disorders) | 1 (1)
Throat pain (General disorders) | 1 (1)
Tinnitus left ear (General disorders) | 1 (1)
Toe pain (General disorders) | 1 (1)
Tongue Lesions (General disorders) | 1 (1)
Tongue Swelling (General disorders) | 1 (1)
Transaminitis (General disorders) | 1 (1)
Upper Extremity Rash (General disorders) | 2 (2)
Upper Extremity Rash * non pruritic* (General disorders) | 1 (1)
Upper GI discomfort (General disorders) | 1 (1)
Urinary Burning (General disorders) | 1 (1)
Urinary Hesitancy (General disorders) | 1 (1)
Vaginal Pruritus (General disorders) | 1 (1)
Vision Changes (General disorders) | 1 (1)
Vitamin D Deficiency (General disorders) | 1 (1)
Vitamin D Insufficiency (General disorders) | 1 (1)
Xerosis (General disorders) | 1 (1)
abdominal cramping (General disorders) | 1 (1)
abdominal rash (General disorders) | 1 (1)
abdominal tenderness (General disorders) | 1 (1)
abdomincal discomfort (General disorders) | 1 (1)
acid reflux (General disorders) | 1 (1)
acute febrile illness (General disorders) | 1 (1)
acute gvhd of skin <25% (General disorders) | 1 (1)
acute liver gvhd (General disorders) | 1 (1)
acute on chronic hyponatremia (General disorders) | 1 (1)
acute renal failure (General disorders) | 1 (1)
agvhd of skin (General disorders) | 1 (1)
anal discomfort (General disorders) | 1 (1)
anion gap acidosis (General disorders) | 1 (1)
ankle pain (General disorders) | 2 (2)
back pruritis (General disorders) | 1 (1)
back rash (General disorders) | 1 (1)
backache (General disorders) | 1 (1)
bilateral ankle edema (General disorders) | 2 (2)
bilateral arm bone pain (General disorders) | 1 (1)
bilateral leg fatigue (General disorders) | 1 (1)
bilateral leg pain (General disorders) | 1 (1)
bilateral lower extremity pain (General disorders) | 2 (2)
bilateral lower leg pain (General disorders) | 1 (1)
bilateral pleural effusion (General disorders) | 1 (1)
bilateral posterior shoulder blade pain (General disorders) | 1 (1)
bilateral subdural hematoma (General disorders) | 1 (1)
black tongue discoloration (General disorders) | 1 (1)
blood blister right upper buccal mucosa (General disorders) | 1 (1)
bloody mucous plug right upper lung (General disorders) | 1 (1)
bone hip pain (General disorders) | 1 (1)
bottom lip pain (General disorders) | 1 (1)
cervical adenopathy (General disorders) | 1 (1)
chest rash (General disorders) | 1 (1)
dry cough (General disorders) | 2 (2)
ecchymosis right arm (General disorders) | 1 (1)
edema bilateral lower extremities (General disorders) | 1 (1)
epigastric discomfort (General disorders) | 1 (1)
epigastric pain (General disorders) | 2 (2)
erythematous rash face (General disorders) | 1 (1)
esophageal NG Tube Trauma (General disorders) | 1 (1)
facial edema (General disorders) | 2 (2)
facial redness (General disorders) | 1 (1)
follicular rash neck (General disorders) | 1 (1)
foot pain (General disorders) | 1 (1)
forehead dryness (General disorders) | 1 (1)
forgetfulness (General disorders) | 1 (1)
hand Tremors (General disorders) | 1 (1)
heart murmur (General disorders) | 1 (1)
heartburn (General disorders) | 5 (5)
hematochezia (General disorders) | 1 (1)
hernia (General disorders) | 1 (1)
hickman Access Complication (General disorders) | 1 (1)
hip pain (General disorders) | 1 (1)
hospital acquired pressure injury to back of neck and sacrum (General disorders) | 1 (1)
hot sensation while urinating (General disorders) | 1 (1)
hypersensitivity right upper chest (General disorders) | 1 (1)
hypogammaglobulinemia (General disorders) | 1 (1)
indigestion (General disorders) | 1 (1)
jaw Pain (General disorders) | 1 (1)
knee effusion (General disorders) | 1 (1)
knee pain (General disorders) | 1 (1)
left Upper extremity Swelling (General disorders) | 1 (1)
left ear lesion (General disorders) | 1 (1)
left eye conjuntiva redness (General disorders) | 1 (1)
left eyelid dryness (General disorders) | 1 (1)
left lower eye lid redness (General disorders) | 1 (1)
left lower eyelid itchiness (General disorders) | 1 (1)
left rib pain (General disorders) | 1 (1)
left sided pleuritic chest pain (General disorders) | 1 (1)
left toe gout (General disorders) | 1 (1)
left wrist swelling (General disorders) | 1 (1)
leg bruising (General disorders) | 1 (1)
leg discomfort (General disorders) | 1 (1)
lesion left lower lip (General disorders) | 1 (1)
lower back pain (General disorders) | 3 (3)
lower extremity Edema (General disorders) | 2 (2)
lower extremity pain (General disorders) | 1 (1)
mental slowing (General disorders) | 1 (1)
mid upper back pain (General disorders) | 1 (1)
migraine (General disorders) | 1 (1)
multifocal pneumonia (General disorders) | 1 (1)
neck discomfort (General disorders) | 1 (1)
neck tightness (General disorders) | 1 (1)
night sweats (General disorders) | 1 (1)
non anion gap metabolic acidosis (General disorders) | 1 (1)
nonocclusive DVT rigiht axillary and basilic veins (General disorders) | 1 (1)
occult blood in stool (General disorders) | 1 (1)
pain at port site (General disorders) | 1 (1)
pain left forearm (General disorders) | 1 (1)
pain right flank (General disorders) | 1 (1)
petechiae bilateral arms (General disorders) | 1 (1)
pruritic Rash Scalp (General disorders) | 1 (1)
pruritic rash back (General disorders) | 1 (1)
pruritic rash face (General disorders) | 1 (1)
rare candida albicans (on BAL) (General disorders) | 1 (1)
rectal irritation (General disorders) | 1 (1)
redness bilateral arms (General disorders) | 1 (1)
respiratory Adenovirus (asymptomatic) (General disorders) | 1 (1)
right ankle pain (General disorders) | 1 (1)
right ankle swelling (General disorders) | 1 (1)
right hand open wound (General disorders) | 1 (1)
right leg cramping (General disorders) | 1 (1)
right pleural effusion (General disorders) | 1 (1)
right posterior thigh pain (General disorders) | 1 (1)
right sided oral gum swelling (General disorders) | 1 (1)
right upper lip ulceration (General disorders) | 1 (1)
scalp discomfort (General disorders) | 1 (1)
scattered rales on bilateral peripheral lungs (General disorders) | 1 (1)
scrotal skin darkening (General disorders) | 1 (1)
shivers (General disorders) | 1 (1)
shortness of breath (General disorders) | 1 (1)
shoulder bruising (General disorders) | 1 (1)
shoulder pain (General disorders) | 2 (2)
skin tear buttock (General disorders) | 1 (1)
sore on lip (General disorders) | 1 (1)
sore throat (General disorders) | 1 (1)
strep viridians ( port culture) (General disorders) | 1 (1)
subconjunctival hemorrhage left eye (General disorders) | 1 (1)
submandibular tenderness (General disorders) | 1 (1)
swelling lower extremities (General disorders) | 1 (1)
throat pain (General disorders) | 4 (4)
trans aminasitis (General disorders) | 1 (1)
tremors bilateral upper extremities (General disorders) | 1 (1)
upper extremity Pruritis (General disorders) | 1 (1)
venoclussive disease (General disorders) | 1 (1)
xerostomia (General disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 2 (2)
BK cystitis (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 2 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
bk viremia positive (Infections and infestations) | 1 (1)
hickman infection (Infections and infestations) | 1 (1)
strepiviridans (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 8 (11)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 24 (26)
Alkaline phosphatase increased (Investigations) | 12 (13)
Aspartate aminotransferase increased (Investigations) | 25 (27)
Blood bilirubin increased (Investigations) | 11 (13)
Blood lactate dehydrogenase increased (Investigations) | 35 (38)
CD4 lymphocytes decreased (Investigations) | 1 (2)
Cardiac troponin I increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 2 (2)
Creatinine increased (Investigations) | 27 (28)
Haptoglobin decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 48 (64)
Neutrophil count decreased (Investigations) | 48 (58)
Platelet count decreased (Investigations) | 55 (65)
Urine output decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 3 (3)
Weight loss (Investigations) | 5 (5)
White blood cell decreased (Investigations) | 51 (66)
Anorexia (Metabolism and nutrition disorders) | 29 (29)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 43 (50)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4)
Hyperlipidemia (Metabolism and nutrition disorders) | 3 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4)
Hyperphosphatemia (Metabolism and nutrition disorders) | 15 (15)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 45 (46)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 46 (47)
Hypocalcemia (Metabolism and nutrition disorders) | 46 (51)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 43 (45)
Hypomagnesemia (Metabolism and nutrition disorders) | 51 (58)
Hyponatremia (Metabolism and nutrition disorders) | 42 (52)
Hypophosphatemia (Metabolism and nutrition disorders) | 35 (35)
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Generalized bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 (12)
Generalized musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain in Knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9)
Worsening muscle/back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vaginal Inclusion Cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 11 (11)
Dysgeusia (Nervous system disorders) | 15 (15)
Headache (Nervous system disorders) | 40 (44)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 10 (11)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 12 (12)
Confusion (Psychiatric disorders) | 4 (4)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 26 (26)
disorientation (Psychiatric disorders) | 1 (1)
word finding difficulties (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Burning while urninating (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 10 (10)
Hematuria (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 12 (13)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4)
Urinary urgency (Renal and urinary disorders) | 1 (1)
urinary hesitancy (Renal and urinary disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pnemonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lip (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Back Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Chest Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis under left eye (Skin and subcutaneous tissue disorders) | 1 (1)
Erhyematous Patches on Back (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythematous Patches bilateral arms (Skin and subcutaneous tissue disorders) | 1 (1)
Erythematous patches bilateral legs (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Facial rash (Skin and subcutaneous tissue disorders) | 2 (2)
ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
Left upper back petechial rash (Skin and subcutaneous tissue disorders) | 1 (1)
Macular Rash Back (Skin and subcutaneous tissue disorders) | 1 (2)
Papular Chest Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Pustular Lesion Right side of nose (Skin and subcutaneous tissue disorders) | 1 (1)
Pustular lesion right side of chin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rash Bilateral Thighs (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Chest (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (11)
Rash upper Extremities (Skin and subcutaneous tissue disorders) | 1 (1)
Skin erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (L) inner cheek (Skin and subcutaneous tissue disorders) | 1 (1)
irritation near seton (Skin and subcutaneous tissue disorders) | 1 (1)
itching (Skin and subcutaneous tissue disorders) | 2 (2)
red spots on hand (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 4 (4)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 28 (29)
Hypotension (Vascular disorders) | 9 (9)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT04339101/Prot_SAP_000.pdf